CLINICAL TRIAL: NCT06671106
Title: Efficacy of an Amine and Zinc Lactate - Containing Mouthrinse in the Home-based Treatment of Plaque-induced Gingivitis in Adolescents. A Single-center, Examiner-blind, Parallel-arm, Randomized Trial
Brief Title: Efficacy of an Amine and Zinc Lactate - Containing Mouthrinse in the Home-based Treatment of Plaque-induced Gingivitis in Adolescents.
Acronym: SPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Collaborators: Consorzio Futuro in Ricerca (Other)
Responsible Party: Principal Investigator, Leonardo Trombelli, Full professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 297-2024-Sper-AUSLFe
Record Dates: First submitted 2024-10-24; First posted 2024-11-04 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Gingivitis
Keywords: mouthrinse; plaque-induced gingivitis; adolescents; oral hygiene; amine lactate; zinc lactate; gingival inflammation; periodontal diseases
MeSH Terms: conditions — Gingivitis; Periodontal Diseases | interventions — Toothbrushing

STUDY DESIGN:
Intervention Model Description: Single center, examiner-blind, parallel-arm, randomized trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Gingivitis - test intervention (Experimental): Gingivitis patients assigned to test intervention will use: manual toothbrush (meridol) and dental floss (meridol) associated with amine and zinc lactate - containing toothpaste (meridol Gum Protection) and amine and zinc lactate - containing mouthrinse (meridol Gum Protection)
  Interventions: Other: toothbrushing; Other: flossing; Device: Toothpaste Product; Device: Mouthrinse
- Gingivitis - control intervention (Active Comparator): Gingivitis patients assigned to control intervention will use: manual toothbrush (meridol) and dental floss (meridol) associated with amine and zinc lactate - containing toothpaste (meridol Gum Protection)
  Interventions: Other: toothbrushing; Other: flossing; Device: Toothpaste Product
- Periodontal health - no treatment (Other): Periodontally healthy subjects will be compared for baseline assessments with gingivitis patients of the other two arms. However, periodontally subjects will conclude their participation in the study within the baseline visit after receiving devices and instructions related to the control intervention.
  Interventions: Other: toothbrushing; Other: flossing; Device: Toothpaste Product

INTERVENTIONS:
Other: toothbrushing — manual toothbrush (meridol)
Other: flossing — dental floss (meridol)
Device: Toothpaste Product — amine and zinc lactate - containing toothpaste (meridol Gum Protection)
Device: Mouthrinse — amine and zinc lactate - containing mouthrinse (meridol Gum Protection)
  Arms: Gingivitis - test intervention

SUMMARY:
The goal of this clinical trial is to evaluate if the adjunctive use of an amine and zinc lactate - containing mouthrinse may give significant benefits in the home-based treatment of plaque-induced gingivitis in adolescents. The study is based on the following hypothesis: the periodontal conditions of participants affected by gingivitis will significantly benefit from the implementation of the self-performed plaque control regimen (consisting of manual toothbrush and amine and zinc lactate toothpaste) with an amine and zinc lactate - containing mouthrinse. The benefit is expected to become manifest in terms of impact on clinical periodontal parameters, ecology of the subgingival environment, patient-reported outcomes and oral-health-related quality of life. In other words, gingivitis participants implementing their self-performed oral hygiene with the investigated mouthrinse are expected to assume a closer profile (based on the outcomes listed above) to periodontally healthy subjects when compared to gingivitis participants not using the investigated mouthrinse.

One hundred fifty participants (100 adolescents with gingivitis and 50 periodontally healthy adolescents) will be selected for the study. Gingivitis patients will be asked to participate in 5 observation intervals: screening visit, study baseline, and 3 follow-up visits (3 weeks, 3 months, 6 months), while periodontally healthy controls will conclude their participation in the study within the baseline visit.

According to the randomization list, at baseline gingivitis patients will receive one of the following home-based oral hygiene regimen:

* test intervention (Gt group): manual toothbrush (meridol) and dental floss (meridol) associated with amine and zinc lactate - containing toothpaste (meridol Gum Protection) and amine and zinc lactate - containing mouthrinse (meridol Gum Protection);
* control intervention (Gc group): manual toothbrush (meridol) and dental floss (meridol) associated with amine and zinc lactate - containing toothpaste (meridol Gum Protection); All periodontally healthy subjects will be assigned control intervention.

At baseline, both gingivitis patients and periodontally healthy subjects will undergo:

* assessment of clinical periodontal parameters;
* subgingival plaque sampling for microbiological analysis;
* assessment of patient-reported outcomes (including oral-health related quality of life) using dedicated questionnaires; Gingivitis subjects will repeat the assessments at 3-week, 3-month, and 6-month follow-up visit.

The 6-month proportion of periodontally healthy participants in each gingivitis group (Gt and Gc) will be regarded as the primary outcome of the study. Changes in clinical parameters, subgingival microbial community profile, and scores related to patient-reported outcomes will be regarded as the secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy;
* eligible for oral care provision by Regional Health Service due to low socio-economic status;
* at least 16 fully erupted teeth (excluding third molars);
* diagnosed with plaque-induced gingivitis (G) or periodontal health (PH) according to the World Workshop case definitions (Trombelli et al. 2018, Chapple et al. 2018);
* willing to participate in the study and capable to fully understand and comply with the study procedures (including questionnaire reading and filling).

Exclusion Criteria:

* pregnant or lactating;
* current smoking;
* motor and/or cognitive deficit impairing compliance with the study intervals or procedures;
* legal guardian not willing to either allow for subject participation in the study or ensure adherence with the study procedures;
* teeth with developmental defects (e.g., enamel pearls/projections);
* untreated oral lesions, including dental caries or endodontic lesions;
* fixed or removable orthodontic appliances or scheduled for orthodontic therapy with a timing not compatible with the experimental phase;
* use of antibiotics in the previous 3 months;
* use of medications that affect the size of the gingival tissues, such as phenytoin, sodium valproate, certain calcium channel-blocking drugs (e.g., nifedipine, verapamil, diltiazem, amlodipine, felodipine), and immune-regulating drugs (e.g., cyclosporine);
* conditions (e.g., Sjögren's syndrome, anxiety, poorly controlled diabetes) or medications (e.g., antihistamines, decongestants, antidepressants) that are associated with hyposalivation.

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-month proportion of periodontally healthy participants | 6 months
  At 6 months, the proportion (range: 0%-100%) of cases of periodontal health (as diagnosed according to the case definition of the 2017 World Workshop) will be evaluated and compared between Gt and Gc groups.

SECONDARY OUTCOMES:
Gingival Index (GI) | 3 weeks, 3 months, 6 months
  GI (without the BoP component) will be assessed on a scale from 0 (no clinically detectable inflammation) to 3 (severe inflammation with spontaneous bleeding) at the mesio-buccal aspects of 6 index teeth (i.e., 1.6, 2.1, 2.4, 3.6, 4.1, 4.4).
  Gt and Gc groups will be compared for the 3-week, 3-month and 6-month changes in Gi.
Plaque score | 3 weeks, 3 months, 6 months
  Plaque score will be evaluated as present (0) or absent (1) at 6 sites (mesio-buccal, buccal, disto- buccal, mesio-lingual, lingual, disto-lingual) of each tooth.
  Gt and Gc groups will be compared for the 3-week, 3-month and 6-month changes in the full-mouth proportion of sites with plaque.
Bleeding on probing (BoP) | 3 weeks, 3 months, 6 months
  BoP will be evaluated as present/absent using a UNC15 probe (Hu-Friedy Italy s.r.l., Milano, Italy) at 6 sites (mesio-buccal, buccal, disto-buccal, mesio- lingual, lingual, disto-lingual) of each tooth.
  Gt and Gc groups will be compared for the 3-week, 3-month and 6-month changes in the full-mouth prevalence of BoP (range: 0%-100%).
Probing depth (PD) | 3 weeks, 3 months, 6 months
  PD will be measured in mm using a UNC15 probe (Hu-Friedy Italy s.r.l., Milano, Italy) at 6 sites (mesio-buccal, buccal, disto-buccal, mesio- lingual, lingual, disto-lingual) of each tooth.
  Gt and Gc groups will be compared for the 3-week, 3-month and 6-month changes in PD.
Clinical attachment level (CAL) | 3 weeks, 3 months, 6 months
  CAL will be measured in mm using a UNC15 probe (Hu-Friedy Italy s.r.l., Milano, Italy) at 6 sites (mesio-buccal, buccal, disto-buccal, mesio- lingual, lingual, disto-lingual) of each tooth.
  Gt and Gc groups will be compared for the 3-week, 3-month and 6-month changes in CAL.
Plaque sampling and microbiological analysis | 3 weeks, 3 months, 6 months
  Plaque sampling will be performed with sterile Mini Five Gracey curettes (Hu-Friedy Italy s.r.l., Milano, Italy) from the subgingival area at the mesio- buccal aspects of 6 index teeth (Manual of Procedures for Human Microbiome Project - Core Microbiome Sampling Protocol Version Number: 12.0; 29 Jul 2010).
  The microbial composition of each sample will be analyzed by a real-time quantitative PCR (qPCR) microarray, providing profiling of microorganisms usually found in dental plaque (Microbial DNA qPCR Array for Oral Disease) (Qiagen, Hilden, Germany). Array assays are designed using the 16S rRNA gene as the target gene and individual primers and hydrolysis-probe detection, increasing specificity of each assay. Amplification will be carried out in a Quant Studio 5 thermocycler (Thermo Fisher Scientific, Milan, Italy), providing simultaneous detection and quantification of 93 different microbial species, including putative and known periodontopathogens.
Patient satisfaction with the use of the oral hygiene regimen | 6 months
  At 6 months, the participant will be asked to state his/her degree of satisfaction with the use of the oral hygiene regimen used during the experimental phase. Satisfaction will be classified as follows: 0- excellent; 1-good; 2- acceptable; 3- poor. The participant will also be asked about possible side effects and complaints related to the use of the assigned products. This evaluation will be performed without the presence of the examiners to enable the participant to give his/her honest opinion.
Oral-health related quality of life (OHrQoL) | Baseline, 6 months
  At baseline and 6 months, participants will be instructed to fill the Child Perceptions Questionnaire for 11- to 14 year-old Children (CPQ11-14). The questionnaire will be filled by the participant under the supervision of the examiner.
  The assessment is developed through 37 questions distributed in 4 sections, which refer to: oral symptoms, functional limitations, emotions related to the condition of the oral cavity, and what role this has in social relationships. Each question will be rated according to the following scale: never (0); once or twice (1); sometimes (2); often (3); every day or almost every day (4).
  The total score will be obtained as the algebraic sum of the single scores, and will range from 0 (indicating no impact of the oral health condition on the quality of life) to 148 (indicating maximum impact of the oral condition on the quality of life).
Adverse events (AEs) | 6 months
  Adverse events will be recorded on a dedicated form, and major adverse events will be immediately communicated to the Operative Unite of Legal Medicine, University - Hospital of Ferrara, Italy.

CONTACTS AND LOCATIONS:
Locations (1):
- Operative Unit of Dentistry, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No
Biological samples (subgingival plaque) will be analyzed at the Section of Microbiology, University of Ferrara, Italy. However, the analysis will be conducted in a blinded fashion (no information related to patient identity and observation interval will be provided for each sample to be analyzed).

REFERENCES:
- [Background] Montesani L, Montesani L, Mateo L, Daep C, Huber N, Isapour G, Zhang YP. Antibacterial and clinical effectiveness of a mouthwash with a novel active system of amine + zinc lactate + fluoride: a randomized controlled trial. Clin Oral Investig. 2024 Jan 13;28(1):90. doi: 10.1007/s00784-023-05487-0. PMID 38217757
- [Background] Trombelli L, Farina R, Silva CO, Tatakis DN. Plaque-induced gingivitis: Case definition and diagnostic considerations. J Clin Periodontol. 2018 Jun;45 Suppl 20:S44-S67. doi: 10.1111/jcpe.12939. PMID 29926492